CLINICAL TRIAL: NCT05143515
Title: The Effectiveness of Physical Activity Calorie Equivalent (PACE) Label on Reducing Food Consumption and Increasing Physical Activity Levels: a Randomized Controlled Trial
Brief Title: The Effectiveness of PACE Label on Reducing Food Consumption and Increasing Physical Activity Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Nuo Zhang, Senior Physical Therapist, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZhangNuo
Record Dates: First submitted 2021-11-09; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACE Label group (Experimental): This group used the PACE label plus calorie label to help participants to know about the number of minutes of walking or running required to burn off the calories in food and drinks.
  Interventions: Behavioral: PACE label
- Calorie Label group (No Intervention): This group used only calorie labels to show the number of calories in food and drinks.

INTERVENTIONS:
Behavioral: PACE label — There were 34 food and drinks choices available for consumption in the pop up café. The labels were displayed next to the food/drink item in the pop up café. The food items were kept in the same position for each participant kitchen to simulate the café environment. Then researchers changed the labels on the display according to the randomisation allocation of each participant. After randomsation participants were informed that they have £10 to spend in the pop-up café and that they could eat the food they selected in a private social eating room.
  Arms: PACE Label group

SUMMARY:
Background: More people are at the risk of chronic disease as the prevalence of obesity increases. It is therefore essential to find ways of helping consumers to make a lower calorie food choice. Current evidence indicates that current food labelling is changing food choices and consumption, but it is of limited effectiveness. Purpose: The purpose of this study is to assess the efficacy of physical activity calorie equivalent (PACE) food labelling on food selection and consumption using a randomised experimental design in pop-up café. Method: This study as a randomised controlled experimental trial (RCT) was conducted in a research kitchen at Loughborough University. Participants were blinded to the exact purpose of the study and randomised to either exposure to PACE labelling plus calorie food labelling or calorie labelling only and asked to select food/drinks for their consumption, in the pop-up café up to a maximum value cost of £10. The study outcomes were the amount of money spent, the number of calories selected, and the amount of food consumed after exposure to the two different types of food labels.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* healthy

Exclusion Criteria:

* allergic to the foods in the pop up café
* chronic disease such as insulin-dependent diabetes
* BMI lower than 16 kg/m2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Money Spent | Immediately after the intervention
  Participants had £10 to spend in the pop-up café and they could eat the food they selected in a private social eating room. The total money they spent were measured when they left the lab.
Calorie Intake | Immediately after the intervention
  The researchers used a digital scale to weigh the original remaining food to the nearest 0.1 gram. The name of food items, the number of calories in each item selected, and the weight of leftover (using calibrated food weighing scales) was recorded for each participant. They were to ensure that all participants had finished eating and left the lab before weighing the remaining food.
The International Physical Activity Questionnaires(IPAQ) | 24 hours after the intervention
  24-hour physical activity questionnaire was sent to them via email one day after the experiment.

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No